CLINICAL TRIAL: NCT05826392
Title: A Single-Session Intervention for Adolescents and Young Adults with Internalizing Problems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Eric A Storch, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-52397
Record Dates: First submitted 2023-03-29; First posted 2023-04-24 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Anxiety; Depressive Symptoms
Keywords: depression; anxiety; growth mindset; neuroplasticity
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Adolescents and young adults (AYA), ages 13-24 will receive a 30-minute, web-based single-session program about growth mindset.
Masking Description: No blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adolescent/Young Adult Self-Administered Web-Based Single-Session Intervention (Experimental): Project Personality is a 30- minute, self-administered, web-based single-session intervention that was developed to help adolescents understand what growth mindsets are and provide them with information about self-changing strategies and coping skills (Schleider & Weisz, 2019). Participants learn about how the brain functions (neuroplasticity), how personality is fluid, and read testimonials from other adolescents about how growth mindsets helped them in school and in their personal lives. Participants also have the opportunity to write notes to other youth, providing them with the advantages of using growth mindsets.
  Interventions: Other: Adolescent/Young Adult Self-Administered Web-Based Single-Session Intervention

INTERVENTIONS:
Other: Adolescent/Young Adult Self-Administered Web-Based Single-Session Intervention — Web-Based, 30-minute self-administered intervention for adolescents
  Other Names: Project Personality

SUMMARY:
With the increasing number of adolescents and young adults (AYA) experiencing depression and anxiety, paired with the lack of time, access, and funding towards social services, AYA need a mental health intervention that is affordable and easily accessible. A single-session intervention (SSI), Project Personality, was developed to improve youth growth mindset and reduce symptoms of internalizing problems, such as anxiety and depression. The purpose of this pilot study is to determine the feasibility of an SSI in adolescents and young adults at a reproductive community health center.

DETAILED DESCRIPTION:
The mental health of adolescents and young adults (AYA) has greatly been impacted since the beginning of the pandemic. With the increasing number of AYA experiencing depression and anxiety, paired with the lack of time, access, and funding towards social services, AYA need a mental health intervention that is affordable and easily accessible. A single-session intervention (SSI) focused on cultivating an AYA's growth mindset has potential to overcome common barriers to care, such as cost, transportation and stigma related to psychological treatment. Furthermore, research shows having a fixed mindset correlate and can predict higher depressive and anxiety symptoms. Teaching adolescents about growth mindsets could decrease the risk of internalizing symptoms. The SSI, Project Personality, was developed to improve youth growth mindset and reduce symptoms of internalizing problems, such as anxiety and depression. The purpose of this pilot study is to determine the feasibility of an SSI in adolescents and young adults at a reproductive community health center.

ELIGIBILITY:
Inclusion Criteria:

* The adolescent or young adult is between the ages of 13 and 24.
* The adolescent or young adult has a score above 5 on either PHQ-9 (Patient Health Questionnaire-9) or GAD-7(General Anxiety Disorder-7).
* The adolescent and their parent participating in the study, or the young adult can read and comprehend English.

Exclusion Criteria:

* The adolescent or the young adult has severe current suicidal/homicidal ideation and/or self-injury requiring medical intervention as defined by the ASQ (Ask Suicide-Screening Questions).
* The adolescent and their parent participating in the study, or the young adult cannot read or comprehend English.
* The adolescent and their parent participating in the study, or the young adult cannot travel to the Baylor College of Medicine (BCM) Teen Health Clinic to receive the single-session intervention.

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Change in Short Mood and Feelings Questionnaire-Child (SMFQ-C) | Baseline (before treatment); 2 weeks post-treatment; 2 months follow-up
  The short version of the self-reported questionnaire that measures depressive symptoms in adolescents 12-17 years old throughout the past 2 weeks. 13 items are scored on a 0-2 scale (0= Not True; 2= True), with a total score between 0-26.
Change in Short Mood and Feelings Questionnaire-Adult (SMFQ-A) | Baseline (before treatment); 2 weeks post-treatment; 2 months follow-up
  The short version of the self-reported questionnaire that measures depressive symptoms in adults throughout the past 2 weeks. 13 items are scored on a 0-2 scale (0= Not True; 2= True), with a total score between 0-26.
Change in PROMIS (Patient-Reported Outcomes Measurement Information System) Anxiety - Child | Baseline (before treatment); 2 weeks post-treatment; 2 months follow-up
  Assesses self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal. 7 items are scored with a total score between 8-40.
Change in PROMIS (Patient-Reported Outcomes Measurement Information System) Anxiety - Adult | Baseline (before treatment); 2 weeks post-treatment; 2 months follow-up
  Assesses self-reported fear, anxious misery, hyperarousal, and somatic symptoms related to arousal in adults. 8 items are scored with a total score between 8-40.

SECONDARY OUTCOMES:
Perceived Primary Control Scale | Baseline (before treatment); 2 weeks post-treatment; 2 months follow-up
  Measures perceived control over academic, social, and behavioral outcomes. Scoring for items 1,2,4,7,9,11,14,15,18,20,22, and 24 are as follows: 0= Very False, 1= Sort of False, 2= Sort of True and 3= Very True. Reverse scoring is needed for items 3,5,6,8,10,12,13,16,17,19,21, and 23 and scoring is as follows: 3= Very False, 2= Sort of False, 1= Sort of True, 0=Very True.
Perceived Secondary Control Scale | Baseline (before treatment); 2 weeks post-treatment; 2 months follow-up
  Measures the ability to adjust oneself to adverse events and how they control their subjective emotional impact. Scoring for items 1,2,5,7,10,14,17,18, and 20 are the following: 0= Very False, 1= Sort of False, 2= Sort of true and 3= Very True. Reverse scoring is needed for items 3,4,6,8,9,11,12,13,16, and 19 and the responses are as follows: 3= Very False, 2= Sort of False, 1= Sort of True, 0= Very True.
The Acceptance and Action Questionnaire-II (AAQ-II) | Baseline (before treatment); 2 weeks post-treatment; 2 months follow-up
  A scale used to evaluate a participant's (young adult) psychological flexibility. 7 items are scored on a 1-7 scale (1= never true; 5 = always true).
Avoidance and Fusion Questionnaire for Youth-8 (AFQ-8) | Baseline (before treatment); 2 weeks post-treatment; 2 months follow-up
  A scale used to evaluate a participant's (adolescent) psychological flexibility. 8 items are scored on a 0-4 scale (0= not at all true; 4 = very true).

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schleider JL, Abel MR, Weisz JR. Do Immediate Gains Predict Long-Term Symptom Change? Findings from a Randomized Trial of a Single-Session Intervention for Youth Anxiety and Depression. Child Psychiatry Hum Dev. 2019 Oct;50(5):868-881. doi: 10.1007/s10578-019-00889-2. PMID 30993499
- [Background] Schleider JL, Dobias M, Sung J, Mumper E, Mullarkey MC. Acceptability and Utility of an Open-Access, Online Single-Session Intervention Platform for Adolescent Mental Health. JMIR Ment Health. 2020 Jun 30;7(6):e20513. doi: 10.2196/20513. PMID 32602846
- See also: with keyword "anxiety" to learn more about anxiety — http://medlineplus.gov/
- See also: with keyword "depression" to learn more about depression — http://medlineplus.gov/genetics/